CLINICAL TRIAL: NCT00814554
Title: PRALIMAP: Effectiveness Evaluation of Three Strategies of Prevention of Overweight and Obesity in Adolescents; a Cluster Randomised Controlled Trial
Brief Title: Effectiveness Evaluation of Three Strategies of Promotion of Healthy Dietary and Physical Activity Behaviours to Prevent Weight Excess Among Teenagers
Acronym: PRALIMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nancy (Other)
Collaborators: National conservatory of arts and crafts (CNAM) (Unknown); Regional institute for health education (IRES) (Unknown); Local school office of the academy of Nancy-Metz (Unknown)
Responsible Party: Briançon Serge Pr, Public Health School - laboratory EA4003
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: pralimap-0610; CNIL-906312; CCTIRS-06.376
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-03

CONDITIONS: Body Weight; Nutrition Processes; Prevention
Keywords: obesity; nutrition; cluster randomized trial; high school; primary prevention
MeSH Terms: conditions — Body Weight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- control (No Intervention): no intervention was carried out in high school
- Educational strategy (Experimental): Educational strategy was carried out in high school.
  Interventions: Behavioral: Educational strategy
- Screening strategy (Experimental): Screening strategy was carried out in high school.
  Interventions: Behavioral: Screening strategy
- Environmental strategy (Experimental): Environmental strategy was carried out in high school.
  Interventions: Other: Environmental strategy
- Educational and Screening strategies (Experimental): Educational strategy and Screening strategy were carried out in high school
  Interventions: Behavioral: Educational strategy; Behavioral: Screening strategy
- Screening and Environmental strategies (Experimental): Screening strategy and Environmental strategy were carried out in high school
  Interventions: Behavioral: Screening strategy; Other: Environmental strategy
- Educational and Environmental strategies (Experimental): Educational strategy and Environmental strategy were carried out in high school
  Interventions: Behavioral: Educational strategy; Other: Environmental strategy
- the three strategies (Experimental): Educational strategy, Screening strategy and Environmental strategy were carried out in high school.
  Interventions: Behavioral: Educational strategy; Behavioral: Screening strategy; Other: Environmental strategy

INTERVENTIONS:
Behavioral: Educational strategy — 1.Educational strategy. The strategy is to implement health promotion actions aiming at developing personal skills to adopt healthy behaviors in the field of nutrition and physical activity in conformity with up-to-date recommendations and references. Each adolescent will be provided with about 50 education hours distributed in individual and collective activities in school (15 hours), interventions during courses (20 hours), and outdoors activities (15 hours).
  Other Names: Axe 1
  Arms: Educational and Environmental strategies; Educational and Screening strategies; Educational strategy; the three strategies
Behavioral: Screening strategy — 2. Screening strategy. Screening includes measurement of BMI and plotting the growing chart with adolescents, measurement of eating troubles. Screening will be performed by the school medical and nurse team. At risk subjects will be defined according to precise criteria and will be referred to the GP and to obesity networks developed by Health Insurance system where they are provided with specific activities with dieticians, physical activity teachers and psychologists. Subjects with psychological difficulties will be referred for psychological care.
  Other Names: Axe 2
  Arms: Educational and Screening strategies; Screening and Environmental strategies; Screening strategy; the three strategies
Other: Environmental strategy — 3. Environmental strategy. The strategy is to develop in schools favorable and supportive environments for healthy behaviors targeting the collective catering and physical activity offer and the establishment policy. Especially actions aim at increase fruits and vegetables availability, water consumption, physical activity inside the schools.
  Other Names: Axe 3
  Arms: Educational and Environmental strategies; Environmental strategy; Screening and Environmental strategies; the three strategies

SUMMARY:
The aim of this study is to compare the effectiveness of three public health intervention strategies to reduce weight excess and obesity prevalence among teenagers within the frame of a public health program aiming at promoting healthy eating and physical activity behaviors.

DETAILED DESCRIPTION:
A cluster randomised trial implemented in 24 high and technical schools including 20 000 fifth-former aims, on a three-year period, at evaluating the effectiveness of three strategies, combined or not, according a 2*2*2 factorial plan, concerning the promotion of healthy dietary and physical activity behaviours: to develop individual skills by individual and collective education, to propose favourable environment, to screen and care for subjects at risk of weight excess. Main outcomes are improvement of knowledge, attitudes and behaviours, mean body mass index (BMI) change, proportion of obese children according to international standards after two years of follow-up, and finally psychological and sociological factors which are facilitators or barriers to such actions. The evidence of the effectiveness of one or the other of the strategies will help to define interventions framework for medical, educative and economic sector actors.

ELIGIBILITY:
Inclusion Criteria:

* Being student in the included public high school in Region of Lorraine (East of France) whatever the age

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5458 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Overweight and obesity according to IOTF references | 0-1-2 years

SECONDARY OUTCOMES:
Knowledge, attitude and behaviors toward nutrition (food and physical activity) | 0-1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Serge Briançon, Pr, Principal Investigator — Public Health School
Locations (1):
- Nancy-University, Vandœuvre-lès-Nancy, France

REFERENCES:
- [Derived] Manneville F, Briancon S, Legrand K, Langlois J, Lecomte E, Omorou AY, Guillemin F. Physical Activity and Eating Behavior Inequalities Mediating the Effects of Socioeconomic Status and Sex on Adolescent Quality of Life: Insights of the PRALIMAP Trial. J Phys Act Health. 2022 Sep 13;19(10):648-657. doi: 10.1123/jpah.2022-0093. Print 2022 Oct 1. PMID 36100207
- [Derived] Langlois J, Omorou AY, Vuillemin A, Briancon S, Lecomte E; PRALIMAP Trial Group. Association of socioeconomic, school-related and family factors and physical activity and sedentary behaviour among adolescents: multilevel analysis of the PRALIMAP trial inclusion data. BMC Public Health. 2017 Feb 8;17(1):175. doi: 10.1186/s12889-017-4070-9. PMID 28178972
- [Derived] Omorou AY, Langlois J, Lecomte E, Vuillemin A, Briancon S; PRALIMAP Trial Group. Adolescents' Physical Activity and Sedentary Behavior: A Pathway in Reducing Overweight and Obesity. The PRALIMAP 2-Year Cluster Randomized Controlled Trial. J Phys Act Health. 2015 May;12(5):628-35. doi: 10.1123/jpah.2014-0035. Epub 2014 Nov 13. PMID 25393601
- [Derived] Bonsergent E, Agrinier N, Thilly N, Tessier S, Legrand K, Lecomte E, Aptel E, Hercberg S, Collin JF, Briancon S; PRALIMAP Trial Group. Overweight and obesity prevention for adolescents: a cluster randomized controlled trial in a school setting. Am J Prev Med. 2013 Jan;44(1):30-9. doi: 10.1016/j.amepre.2012.09.055. PMID 23253647
- [Derived] Legrand K, Bonsergent E, Latarche C, Empereur F, Collin JF, Lecomte E, Aptel E, Thilly N, Briancon S. Intervention dose estimation in health promotion programmes: a framework and a tool. Application to the diet and physical activity promotion PRALIMAP trial. BMC Med Res Methodol. 2012 Sep 19;12:146. doi: 10.1186/1471-2288-12-146. PMID 22992391
- [Derived] Briancon S, Bonsergent E, Agrinier N, Tessier S, Legrand K, Lecomte E, Aptel E, Hercberg S, Collin JF; PRALIMAP Trial Group. PRALIMAP: study protocol for a high school-based, factorial cluster randomised interventional trial of three overweight and obesity prevention strategies. Trials. 2010 Dec 6;11:119. doi: 10.1186/1745-6215-11-119. PMID 21134278